CLINICAL TRIAL: NCT07002918
Title: The Impact of Paraspinal Muscle Atrophy in Lumbar Spinal Fusion Outcomes
Brief Title: The Impact of Paraspinal Muscle Atrophy in Spine Surgeries
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Adnan Ahmad Elkamel, Resident Doctor, Assiut University
Other Study IDs: Paraspinal muscle atrophy
Record Dates: First submitted 2025-05-25; First posted 2025-06-04 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Paraspinal Muscles; Degenerative Lumbar Diseases
Keywords: paraspinal muscles atrophy; Degenerative lumbar spine diseases; lumbar spine fusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to learn about the role of pre-operative paraspinal muscle atrophy in outcomes of lumbar spine fusion surgeries in patients with degenerative lumbar spine diseases. The main question it aims to answer is:

Does paraspinal muscle atrophy worsen lumbar spine fusion surgeries outcomes? Participants undergoing lumbar spine fusion surgeries as part of their treatment for degenerative lumbar spine diseases will answer survey questions about their low back pain and daily activities for 1 year.

DETAILED DESCRIPTION:
Lumbar spine fusion surgery is a widely performed intervention worldwide with the rate steadily increasing. This trend reflects the growing burden of degenerative spinal disorders (DSD) and low back pain (LBP), which globally affect an estimated 266 million individuals (3.63% of the global population) each year. Socioeconomic factors are important risk aspects for lumbar pain and disability both directly and indirectly. Despite the widespread use of lumbar fusion surgery, outcomes are not uniformly successful. A significant proportion of patients experience poor postoperative results, with studies indicating that 33% of patients report treatment failure, including a 22% worsening rate after surgery for lumbar spinal stenosis. Factors associated with these poor outcomes include prolonged back pain duration (>12 months), prior spinal surgery, and advanced age (>70 years). One critical yet often overlooked factor contributing to poor outcomes is paraspinal muscle atrophy. The paraspinal muscles and vertebrae are interdependent tissues, and the health of these muscles plays a vital role in spinal stability and function. The multifidi, erector spinae, psoas, and quadratus lumborum muscles provide support for the lower back. Numerous studies have explored the degeneration or atrophy of back muscles and the reduction in back extensor muscle strength in patients with lower back pain. Patients with high lumbar muscularity and mild fatty infiltration ratio observed on preoperative MRI demonstrated more promising clinical and radiographic outcomes after lumbar interbody fusion. As the prevalence of degenerative spinal conditions continues to rise globally, understanding the role of paraspinal muscle health in surgical success is critical. By prioritizing patient selection based on modifiable risk factors, clinicians can enhance postoperative outcomes and mitigate the economic and clinical burdens associated with lumbar fusion surgery.

* Sample Size Calculation:

Based on determining the main outcome variable, The estimated minimum required sample size is 55 patients.

The sample size was calculated using Epi-info version 7 software, based on the following assumptions:

Main outcome variable is to determine the impact of paraspinal muscle atrophy on lumbar spine fusion outcomes. Previous studies indicate a significant decrease in paraspinal muscle volume one year after surgery, dropping from 67.8% to 60.4%. This reduction correlates significantly with physical and mental outcomes, as well as pain levels. With 80% confidence, the margin of error for these findings is estimated to be within 3%.

- Study tools (in detail, e.g., lab methods, instruments, steps, chemicals, …):

A. Preoperative:

* Magnetic resonance imaging (MRI) of lumbar spine will be used to measure the total cross-sectional area (TCSA), functional cross-sectional area (FCSA) and fatty infiltration (FI) of erector spinae (ES), multifidus (MF) and psoas major (PM) at the level of diseased segment together with one level above & below using ImageJ software v1.54p.
* plain X-rays will be used to measure local kyphotic angle and lumbar lordosis using Surgimap software v2.3.2.1.
* Oswerty disability index Arabic version (ODI)
* EuroQol-5-dimension 5-level Arabic version (EQ-5D-5L)
* Visual analogue scale (VAS) B. Day one postoperative: Postoperative X-ray. C. Two weeks postoperative: Wound check. ODI, EQ-5D-5L, Visual Analogue Score. D. Six weeks postoperative: Wound check. ODI, EQ-5D-5L, Visual Analogue Score. E. Three months postoperative: ODI, EQ-5D-5L, Visual Analogue Score. F. Six months Postoperative: ODI, EQ-5D-5L, Visual Analogue Score, X-ray. G. One year Postoperative: ODI, EQ-5D-5L, Visual Analogue Score, X-ray, MRI if the patient is still complaining.

ELIGIBILITY:
Inclusion Criteria:

* Patients with degenerative lumbar spine diseases undergoing lumbar spinal fusion.

Exclusion Criteria:

* Long-level fusion ≥ 3 levels.
* History of previous lumbar surgery.
* Patients diagnosed with spondylolysis.
* Other pathological conditions such as fractures, infections or tumors.
* Uncontrolled comorbidities.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing lumbar spinal fusion at Assiut University Hospitals, Department of Orthopedic surgery and Traumatology.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Oswerty disability index Arabic version (ODI) | Baseline, 2 weeks postoperative, 6 weeks postoperative, 3 months postoperative, 6 months postoperative and 1 year postoperative.
  The Oswestry Disability Index (ODI) translates low back pain disability into a numerical score for better understanding and communication. It's a questionnaire used to assess the impact of low back pain on a person's daily life, work, and ability to perform specific tasks. The ODI translates into a score from 0-100, with higher scores indicating greater disability. This score helps clinicians and researchers quantify the functional disability caused by low back pain.

SECONDARY OUTCOMES:
Visual analogue scale (VAS) | Baseline, 2 weeks postoperative, 6 weeks postoperative, 3 months postoperative, 6 months postoperative and 1 year postoperative.
  A Visual Analogue Scale (VAS) is a measurement tool used to assess subjective experiences like pain or discomfort by having a person mark a point on a continuous line representing the range from "no pain" to "worst imaginable pain". Zero is equivalent to no pain and 10 indicates the worst possible pain.
Local kyphotic angle | Baseline, 1 day postoperative, 6 months postoperative and 1 year postoperative.
  In the context of degenerative spine disease, the local kyphotic angle refers to the increased forward curvature (kyphosis) at a specific level of the spine, often between two adjacent vertebral bodies. This local kyphosis can result from various factors, including vertebral collapse, disc degeneration, or changes in vertebral shape associated with aging. The local kyphotic angle is typically measured using X-ray images, with the angle formed by the upper and lower endplates of the vertebral bodies.
Lumbar lordosis | Baseline, 1 day postoperative, 6 months postoperative and 1 year postoperative.
  In degenerative lumbar spine disease, the normal inward curve of the lower back (lumbar lordosis) can change. This change can manifest as a loss of lordosis (flattening of the curve) or an increase in lordosis (excessive curve). It is measured using X-rays of lateral view of lumbar spine by using the lumbosacral angle (LSA), which is the angle between the top of L1 (the first lumbar vertebra) and the top of the sacrum. The Cobb angle method, using lines drawn along the superior endplates of L1 and S1.
EuroQol-5-dimension 5-level Arabic version (EQ-5D-5L) | Baseline, 2 weeks postoperative, 6 weeks postoperative, 3 months postoperative, 6 months postoperative and 1 year postoperative.
  The EuroQol 5-Dimension 5-Level (EQ-5D-5L) questionnaire measures health-related quality of life by assessing five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression, each with five levels of severity. These levels range from "no problems" to "extreme problems" and the responses are combined to create a unique health state profile.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed S Abdelgawaad, Professor Doctor, Study Chair — Assiut University; Amr H Ahmed, MD, Study Director — Assiut University; Adnan A Elkamel, Bachelor degree, Principal Investigator — Assiut University
Locations (1):
- Assiut University, Asyut, Asyut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Shawky Abdelgawaad A, El-Sharkawi M, Sarhan AM, Hassanien MA, Aziz M. Validation of the arabic version of the EuroQol-5-dimension 5-level (EQ-5D-5 L) in patients with spinal degenerative diseases. BMC Public Health. 2024 Apr 23;24(1):1119. doi: 10.1186/s12889-024-18367-3. PMID 38654180
- [Background] Algarni AS, Ghorbel S, Jones JG, Guermazi M. Validation of an Arabic version of the Oswestry index in Saudi Arabia. Ann Phys Rehabil Med. 2014 Dec;57(9-10):653-63. doi: 10.1016/j.rehab.2014.06.006. Epub 2014 Aug 4. PMID 25262247
- [Background] Waschke A, Hartmann C, Walter J, Dunisch P, Wahnschaff F, Kalff R, Ewald C. Denervation and atrophy of paraspinal muscles after open lumbar interbody fusion is associated with clinical outcome--electromyographic and CT-volumetric investigation of 30 patients. Acta Neurochir (Wien). 2014 Feb;156(2):235-44. doi: 10.1007/s00701-013-1981-9. Epub 2014 Jan 3. PMID 24384989
- [Background] Mayer TG, Vanharanta H, Gatchel RJ, Mooney V, Barnes D, Judge L, Smith S, Terry A. Comparison of CT scan muscle measurements and isokinetic trunk strength in postoperative patients. Spine (Phila Pa 1976). 1989 Jan;14(1):33-6. doi: 10.1097/00007632-198901000-00006. PMID 2913665
- [Background] Cooper RG, St Clair Forbes W, Jayson MI. Radiographic demonstration of paraspinal muscle wasting in patients with chronic low back pain. Br J Rheumatol. 1992 Jun;31(6):389-94. doi: 10.1093/rheumatology/31.6.389. PMID 1534505
- [Background] You KH, Cho M, Lee JH. Effect of Muscularity and Fatty Infiltration of Paraspinal Muscles on Outcome of Lumbar Interbody Fusion. J Korean Med Sci. 2023 May 22;38(20):e151. doi: 10.3346/jkms.2023.38.e151. PMID 37218352
- [Background] Alhaug OK, Dolatowski FC, Solberg TK, Lonne G. Predictors for failure after surgery for lumbar spinal stenosis: a prospective observational study. Spine J. 2023 Feb;23(2):261-270. doi: 10.1016/j.spinee.2022.10.010. Epub 2022 Nov 5. PMID 36343913
- [Background] Sihvonen T, Herno A, Paljarvi L, Airaksinen O, Partanen J, Tapaninaho A. Local denervation atrophy of paraspinal muscles in postoperative failed back syndrome. Spine (Phila Pa 1976). 1993 Apr;18(5):575-81. doi: 10.1097/00007632-199304000-00009. PMID 8484148
- [Background] Ravindra VM, Senglaub SS, Rattani A, Dewan MC, Hartl R, Bisson E, Park KB, Shrime MG. Degenerative Lumbar Spine Disease: Estimating Global Incidence and Worldwide Volume. Global Spine J. 2018 Dec;8(8):784-794. doi: 10.1177/2192568218770769. Epub 2018 Apr 24. PMID 30560029